CLINICAL TRIAL: NCT04530942
Title: The Efficacy and Prediction of Deep Brain Stimulation for Treatment-resistant Depression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Bomin Sun, Principal Investigator, Ruijin Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2020 DBS for TRD
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Major Depressive Disorder; Deep Brain Stimulation
Keywords: Treatment Resistant Depression; Deep Brain Stimulation; Ventral Capsule/Ventral Striatum
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Intervention Model Description: The study starts with a longitudinal open-label phase followed by a randomized, double blind crossover phase. In the crossover phase, patients are randomized to active DBS for 2 weeks, followed by sham DBS for 2 weeks, or vice versa. The patients' post-surgery duration need to be more than 6 months when they entered the randomized cross-over phase.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active DBS then Sham DBS (Experimental): After more than 6 months open-lable period, some patients will take DBS ON for two weeks with the optimal stimulation parameters and then take DBS OFF for two weeks.
  Interventions: Device: Deep brain stimulation(Active); Device: Deep brain stimulation(Sham)
- Sham DBS then Active DBS (Experimental): After more than 6 months open-lable period, some patients will take DBS OFF for two weeks and then take DBS ON for two weeks with the optimal stimulation parameters.
  Interventions: Device: Deep brain stimulation(Active); Device: Deep brain stimulation(Sham)

INTERVENTIONS:
Device: Deep brain stimulation(Active) — DBS On with the optiomal parameters
  Other Names: DBS On
Device: Deep brain stimulation(Sham) — DBS On with 0V Amplitude
  Other Names: DBS Off

SUMMARY:
Several open-label trials have shown the therapeutic promise of deep brain stimulation (DBS) targeted to striatal and surrounding capsular areas in treatment-resistant depression (TRD). However, the results of placebo-controlled trials have been mixed, with one showing a large difference between active and sham DBS and another finding no difference.

Main aim of this study is establishing whether active DBS results in more treatment responders than sham DBS. Secondary aims are establishing an adverse events profile, establishing effects on quality of life,neuropsychological and neuroimaging measures, and finding predictors of response.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is a highly prevalent psychiatric disorder, with an estimated lifetime prevalence of 14.6% across high-income countries.Effective therapeutic options for MDD include psychotherapy, different classes of antidepressants, and electroconvulsive therapy (ECT). Nevertheless, up to 30% of patients do not respond to four consecutive antidepressant strategies and 52% of pharmacotherapy resistant patients do not respond to ECT.Such patients are designated an advanced stage of Treatment Resistant Depression (TRD), which is associated with more hospitalizations, more suicide attempts, and higher costs than non-TRD patients.

Deep Brain Stimulation (DBS) is a promising therapeutic option for TRD patients. DBS consists of implanting electrodes in specific brain areas and then optimizing stimulation parameters (e.g. voltage, frequency, pulse width) to modulate brain activity of the targeted area. Since 2005, several open label trials have reported promising effects of DBS in TRD, targeting different brain structures involved in the neurobiology of MDD: the Subcallosal Cingulate Gyrus (SCG),Medial Forebrain Bundle (MFB),Ventral Capsule/Ventral Striatum (VC/VS), and Nucleus Accumbens (NAc). Response rates, defined as a symptom decrease of at least 50%, range from 30% to 90% with most studies finding a response rate around 50%.

However, results of the first two randomized trials are mixed. The first randomized, controlled trial (RCT) of VC/VS DBS in TRD did not find differences in response rates following active (3 of 14 patients) or sham stimulation (2 of 15 patients) after four months of stimulation. In contrast, another group found a strong antidepressant effect in 16 patients with TRD following active ventral Anterior Limb of the Internal Capsule (vALIC) DBS compared to sham stimulation in a randomized crossover phase.

Therefore, this trial aims to establishing whether active DBS results in more treatment responders than sham DBS. Secondary aims are establishing an adverse events profile, establishing effects on quality of life,neuropsychological and neuroimaging measures, and finding predictors of response.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis: Major Depressive Disorder according to the ICD-10 criteria based on a psychiatric interview
* Age: 18-65 years old
* HAMD-17 total ≥17
* Chronic illness with current episode ≥ 24 months duration and/or Illness with at least a total of 4 lifetime episodes (including current episode≥ 12 months) and a minimum of 5 years since the onset of the first depressive episode
* Treatment refractory defined as failure of: at least 3 adequate treatments from at least two distinctly different classes (SSRI, SNRI, NaSSA, TCA +, lithium-addition) for a period of 6-8 weeks or more weeks. Adequate psychotherapy. At least 1 session of ECT, for which the series of ECT was terminated either due to adverse effects or insufficient response (including at least 6 sessions of bilateral ECT); unavailable, rejective or intolerable to ECT
* remain stable with the current anti-depressive medicine for the last month
* Able and willing to give written informed consent
* Able to fully understand the consequences of the procedure

Exclusion Criteria:

* Schizophrenia /history of psychosis unrelated to MDD
* Severe personality disorder (assessed by SCID-II)
* Abnormal brain MRI
* Neurological disease (e.g., Parkinson's disease)
* Previous sterosurgery
* Any medical contraindication to surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
the comparison between the Hamilton Depression Scale(HAMD-17) scores after active and sham phase | Baseline (preoperative),one month, 3 months, 6 months, 6.25 months, 6.5 months, 9 months, 12 months, 18months
  Effect size of comparison between HAMD-17 scores at two weeks when the active and sham phase end. The score of HAMD-17 ranges from 0 to 50. Higher HAMD-17 score indicates more severe depression.

SECONDARY OUTCOMES:
changes in the Montgomery-Asberg Depression Rating Scale(MADRS) | Baseline (preoperative),one month, 3 months, 6 months, 6.25 months, 6.5 months, 9 months, 12 months, 18months
  Effect size of active compared to sham stimulation score before and after the sham and treatment periods. The score of the scale ranges from 0 to 60. Higher MADRS score indicates more severe depression.
changes in the Quick Inventory of Depression Scale(QIDS-SR16) | Baseline (preoperative),one month, 3 months, 6 months, 6.25 months, 6.5 months, 9 months, 12 months, 18months
  Effect size of active compared to sham stimulation score before and after the sham and treatment periods. The score of the scale ranges from 0 to 42. Higher QIDS-SR16 score indicates more severe depression.
changes in the Depression and Somatic Symptoms Scale(DSSS) | Baseline (preoperative),one month, 3 months, 6 months, 6.25 months, 6.5 months, 9 months, 12 months, 18months
  Effect size of active compared to sham stimulation score before and after the sham and treatment periods. The score of the scale ranges from 0 to 66. Higher DSSS score indicates more severe depression and anxiety.
changes in the Dimensional Anhedonia Rating Scale(DARS) | Baseline (preoperative),one month, 3 months, 6 months, 6.25 months, 6.5 months, 9 months, 12 months, 18months
  DARS is a self-reported dynamic scale that measures desire, motivation, effort and consummatory pleasure across hedonic domains. Higher scores indicate lower degrees of anhedonia.
changes in Hamilton Anxiety Scales(HAMA) | Baseline (preoperative),one month, 3 months, 6 months, 6.25 months, 6.5 months, 9 months, 12 months, 18months
  Clinician administered assessment.The score of the scale ranges from 0 to 56. The higher scores means more severe anxiety.
changes in World Health Organization Quality of Life-BREF(WHO-BREF) | Baseline (preoperative),one month, 3 months, 6 months, 6.25 months, 6.5 months, 9 months, 12 months, 18months
  The World Health Organization Quality of Life - BREF (WHOQOL-BREF) is a self report questionnaire which assesses 4 domains of quality of life (QOL): physical health, psychological health, social relationships, and environment. It contains 26 items which is a 5 points scale. The higher score means better quality of life.
changes in the MOS item short from health survey (SF-36) | Baseline (preoperative),one month, 3 months, 6 months, 6.25 months, 6.5 months, 9 months, 12 months, 18months
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and are now widely utilized by managed care organizations and by Medicare for routine monitoring and assessment of care outcomes in adult patients. The higher score means better quality of life.
changes in Sheehan Disability Scale | Baseline (preoperative),one month, 3 months, 6 months, 6.25 months, 6.5 months, 9 months, 12 months, 18months
  Self-rating scale. The SDS is a composite of three self-rated items designed to measure the extent to which three major domains in the patient's life are functionally impaired by psychiatric or medical symptoms. The SDS assesses functional impairment in three major life domains: work, social life/leisure activities, and family life/home responsibilities. The higher scores mean more severity of disability.
changes in Neuropsychological measures(Scores of Thinc-it tasks) | Baseline (preoperative), 6.25 months, 6.5 months, 18months
  Neuropsychological measures contains six domains of cognition which are episodic memory, working memory,attention, executive functions, psychomotor speed and social cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Bomin Sun, PhD, Principal Investigator — Ruijin Hospital
Locations (1):
- Functional neurosurgery of Shanghai Jiaotong University affiliated Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dougherty DD, Rezai AR, Carpenter LL, Howland RH, Bhati MT, O'Reardon JP, Eskandar EN, Baltuch GH, Machado AD, Kondziolka D, Cusin C, Evans KC, Price LH, Jacobs K, Pandya M, Denko T, Tyrka AR, Brelje T, Deckersbach T, Kubu C, Malone DA Jr. A Randomized Sham-Controlled Trial of Deep Brain Stimulation of the Ventral Capsule/Ventral Striatum for Chronic Treatment-Resistant Depression. Biol Psychiatry. 2015 Aug 15;78(4):240-8. doi: 10.1016/j.biopsych.2014.11.023. Epub 2014 Dec 13. PMID 25726497
- [Background] Bergfeld IO, Mantione M, Hoogendoorn ML, Ruhe HG, Notten P, van Laarhoven J, Visser I, Figee M, de Kwaasteniet BP, Horst F, Schene AH, van den Munckhof P, Beute G, Schuurman R, Denys D. Deep Brain Stimulation of the Ventral Anterior Limb of the Internal Capsule for Treatment-Resistant Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2016 May 1;73(5):456-64. doi: 10.1001/jamapsychiatry.2016.0152. PMID 27049915
- [Background] Dandekar MP, Fenoy AJ, Carvalho AF, Soares JC, Quevedo J. Deep brain stimulation for treatment-resistant depression: an integrative review of preclinical and clinical findings and translational implications. Mol Psychiatry. 2018 May;23(5):1094-1112. doi: 10.1038/mp.2018.2. Epub 2018 Feb 27. PMID 29483673
- [Derived] Wang L, Zhang Y, Wang Y, Ding Q, Dai L, Hu K, Ye K, Lv X, Zhang X, Mandali A, Manssuer L, Sonkusare S, Zhao Y, Huang P, Qiu X, Pan Y, Lai Y, Li D, Liu W, Zhan S, Sun B, Voon V. Prefrontal-bed nucleus of the stria terminalis physiological and neuropsychological biomarkers predict therapeutic outcomes in depression. Nat Commun. 2025 Nov 18;16(1):10034. doi: 10.1038/s41467-025-65179-z. PMID 41253805